CLINICAL TRIAL: NCT01425827
Title: Duloxetine for Pain in Older Adults With Knee Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, Professor of Rheumatology, University of Alexandria
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: alexmed116619163
Record Dates: First submitted 2011-08-19; First posted 2011-08-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pain Reduction; Function Improvement
Keywords: duloxetine; osteoarthritis; pain; function
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: duloxetine HCL — 60 mg/day duloxetine for 16 weeks
Drug: placebo — similar looking tablets to the active agent for 16 weeks

SUMMARY:
Osteoarthritis (OA), a common disabling condition, is the commonest type of arthritis worldwide.Pain is the leading symptom and is often chronic in na. Current treatment options have had limited symptomatic effect and are associated with significant side effects. Duloxetine, a selective serotonin norepinephrine reuptake inhibitor has been demonstrated to have, besides its antidepressant properties, a centrally acting analgesic effect.

The aim of the present study was to investigate the efficacy of duloxetine in reducing pain in older adults with knee OA.

288 patients aged 65 years and above with ACR clinical and radiographic criteria of primary knee OA attending the outpatient clinic of our institution were enrolled in this study. All patients underwent a physical examination and where questioned about the number of flares. Exclusion criteria included any inflammatory, autoimmune, psychiatric illness and morbid obesity. Patients were randomized 1:1. One hundred and forty four received 60mg/day of duloxetine HCL and 144 received placebo together with their usual therapy for 16 weeks. The primary outcome measure was pain reduction. Secondary outcome measures included improvements in physical functioning scores. Pain was assessed using the Brief Pain Inventory (BPI) and Visual Analogue pain Scale, (VAS, 0-100 mm). Functional assessment using the self-reported physical function as measured with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), WOMAC pain and stiffness scores and the Geriatric Depression Scale (GDS) was conducted. Alterations in dosage of analgesic/NSAID drugs used were recorded. Safety and tolerability were also assessed. Data was collected at baseline and at monthly intervals for 4 months. All staff involved in data collection was blinded to the treatment assignment groups.

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis

Exclusion Criteria:

* inflammatory conditions
* autoimmune disorders
* psychiatric illness
* morbid obesity

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anna Abou-Raya, MD, Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt

REFERENCES:
- [Derived] Abou-Raya S, Abou-Raya A, Helmii M. Duloxetine for the management of pain in older adults with knee osteoarthritis: randomised placebo-controlled trial. Age Ageing. 2012 Sep;41(5):646-52. doi: 10.1093/ageing/afs072. Epub 2012 Jun 27. PMID 22743149